CLINICAL TRIAL: NCT03643198
Title: Oral Antibiotics for Anal Abscess to Diminish the Developement of Perianal Fistula
Brief Title: Oral Antibiotics for Anal Abscess
Acronym: OFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, David Parés MD, PhD, David parés. MD, PhD. Consultant Surgeon. Associate professor, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-001-bcn.nord
Record Dates: First submitted 2018-08-19; First posted 2018-08-22 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Anal Fistula; Anal Abscess
MeSH Terms: conditions — Rectal Fistula | interventions — Anti-Bacterial Agents; Metronidazole; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: 2 arms
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL (Sham Comparator): The control group will receive two types of placebo tablets that look identical to Ciprofloxacin and Metronidazole respectively, with similar doses and frequencies.
  Interventions: Other: CONTROL
- TREATMENT (Active Comparator): In the study group, patients will receive oral treatment with Ciprofloxacin at a dose of 500 mg every 12 hours and Metronidazole 500 mg every 8 hours for a period of 7 days.
  Interventions: Drug: ANTIBIOTIC (METRONIDAZOLE AND CIPROFLOXACIN); Other: CONTROL

INTERVENTIONS:
Drug: ANTIBIOTIC (METRONIDAZOLE AND CIPROFLOXACIN) — The control group will receive two types of placebo tablets that look identical to Ciprofloxacin and Metronidazole respectively, with similar doses and frequencies.
  Arms: TREATMENT
Other: CONTROL — NO treatment

SUMMARY:
BACKGROUND Anal abscess and perianal fistula is a high prevalence disorder in general population that affect adult patients on young ages, affecting them significantly their social and quality of life. There is clinical evidence that the origin of most perianal fistulas (60%) is with an episode one year before of a perianal abscess. In fact, the established cryptoglandular hypothesis considered the origin of anal fistula, a chronic infectious disease starting on a clinical episode of an anal glands abscess. However, controversy exists regarding the role of antibiotics in the development of anal fistula after incision and drainage of perianal abscess. Nowadays, only two single-centre randomized controlled trials has been published addressing this issue, with inconclusive results. The MAIN OBJECTIVE of the study is to examine the clinical benefit of antibiotic therapy in patients with a perianal abscess, to avoid the development of a perianal fistula. METHODOLOGY We designed a prospective, multicentre double-blind placebo trial to analyse the clinical benefit of a course of antibiotics after perianal abscess drainage to diminish the probability of development of perianal fistula in the follow up of patients. Patients with anal abscess will be allocated randomly either to receive 7 days of oral metronidazole/ciprofloxacin in addition to their standard care or to receive standard care and placebo, after they will be discharged from the hospital. Patients will be followed clinically at different intervals during one year in order to know if they develop anal fistula. Also a quality of life assessment at the end of the study will be evaluated. EXPECTED RESULTS We expected that patients allocated to antibiotic treatment would develop a significant less anal fistulas in their follow-up with a related significant better quality of life. Thus, a change on standard of care led by our group, may be achieved.

DETAILED DESCRIPTION:
METHODS This project is a 3-year study.

Trial Design:

This is a multicentre, double-blind placebo trial to investigate the effect of oral antibiotics after anal abscess drainage to diminish the development of an anal fistul.

This Clinical Trial will consist of two parallel study groups with a (1:1) randomization, masking by double-blind technique and placebo control.

Participants:

The participants of this study will be eligible among those who will be attended on the emergency department of each participant hospital during inclusion period.

Interventions:

This study will include patients who come to the emergency room due to perianal abscesses and who will be incised and drained of the lesion by local anaesthesia (in emergency boxes) or by regional or general anaesthesia (in the operating room). A standard procedure will be followed with draining the purulent contents and then instilling a solution composed of saline and iodine through the wound; as well as manual exploration and lysis of intracavity septa.

In all cases as it it standardized, the wound will be left open with insinuated gauze or a latex drainage (Penrose) when necessary.

The patients, once selected, will be randomly distributed (by specific software) in two parallel groups, in one of which the intervention will be evaluated. In the study group, patients will receive oral treatment with Ciprofloxacin at a dose of 500 mg every 12 hours and Metronidazole 500 mg every 8 hours for a period of 7 days. The control group will receive two types of placebo tablets that look identical to Ciprofloxacin and Metronidazole respectively, with similar doses and frequencies.

Postoperative controls and follow-up will be carried out at 1, 3, 6 and 12 months after treatment and will include an endoanal ultrasound (US) at 6 months.

Studied variables:

The following variables will be analysed:

* Epidemiological variables: Age, gender.
* Smoking status
* Comorbidities
* Obesity (Body Mass Index)
* Cultures of abscess
* Characteristics of anal abscess: Location, type of drainage.
* Selected arm: Group treatment (antibiotics) vs. Control group (placebo)
* Clinical follow up (anal fistula or not) at 1, 3, 6 and 12 months.

The diagnosis of anal fistula is standarized by specialist in General Surgery.

* Type of anal fistula developed
* Endoanal US at 6 months
* Adverse events of treatment
* Quality of life (general health with SF-36 test and an specific test related to quality of life in patients with anal fistula, both tests validated to Spanish language) at 12 months (end of follow up)

Expected outcomes:

Once the patients with diagnosis of perianal abscess treated with incision and drainage were included, the objective of our study will be to evaluate the proportion of patients who developed perianal fistula between the two study groups (with oral antibiotics and with placebo). It will be recorded as the presence of a perianal fistula when the participants present a history of symptoms compatible with it, as well as the existence of a communication between the perianal cutaneous tissue and the anal canal during the clinical examination performed or even evidenced in the endoanal ultrasound during the controls that will be carried out up to 12 months after the intervention. For better evaluation and registration abscesses will be classified according to their complexity: subcutaneous, intersphincteric, ischiorectal and according to their anatomical location: anterior, posterior, lateral, right and left. These data will be collected at the time of the surgical exploration during the initial treatment with incision and drainage.

Fistulas will be classified by Parks classification in the following: subcutaneous, intersphinterian, transphincteric, suprasphinteric, extraphincteric. These data will be collected at the time of the clinical examination during the controls.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years old
* Clinical diagnosis of perianal abscess

Exclusion Criteria:

* Participants who have a history of previous perianal abscesses.
* Inflammatory bowel disease
* Patients who already have a perianal fistula
* Patients with perianal cancer and / or pelvic radiotherapy
* Perianal trauma
* Immunodeficiency
* Diabetes
* Pregnancy or lactation
* Valvular heart disease or prosthetic valve carriers
* Spontaneous drainage
* Previous use of antibiotics
* Patients with a known allergy to Ciprofloxacin or Metronidazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Perianal fistula incidence | 12 months
  Formation of perianal/anal fistula at follow-up during 12 months after anal abscess. This outcome will be defined clinically and with anal ultrasound.

SECONDARY OUTCOMES:
Improving on Quality of life | 12 months
  Measurement of quality of life. We will use the test named SF36 in its Validated version in Spanish. This test evaluates the health-related quality of life with answers of 36 questions and punctuates from 0 to 100, being 100 the maximum score (Better quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- David Parés, Barcelona, Spain